CLINICAL TRIAL: NCT05745493
Title: Promoting Social Connection to Prevent Late-Life Suicide
Brief Title: Study 1: Social Engage Coaching R61 Phase
Acronym: R61 Phase
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kimberly Van Orden, Associate Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 408656; R61MH129476 (NIH)
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Social Isolation; Loneliness; Suicide Ideation; Quality of Life
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social Engage Coaching (S-ENG) (Experimental): Social Engage Coaching is 10 individual sessions of coaching to increase social connection.
  Interventions: Behavioral: Social Engage Coaching (S-ENG)

INTERVENTIONS:
Behavioral: Social Engage Coaching (S-ENG) — Social Engage Coaching (S-ENG) involves 10 individual coaching sessions focused on increasing social connection. S-ENG is a stepped, modular intervention that was developed to allow personalization to a given subject's needs, preferences, and individualized barriers to social connection. Early sessions include psychoeducation on the importance of social connection; a values clarification exercise on aspects of connection most important to subjects; and assessment of current social networks and social activities. Together, the coach and subject create a conceptualization of reasons for loneliness and identify personalized activities most likely to impact loneliness. The primary activity is 'action planning,' which involves selecting a social goal for the week, brainstorming ways to meet the goal, identifying barriers, and selecting specific actions to take before the next session. The first 8 sessions are offered weekly and the final two are monthly booster sessions.

SUMMARY:
The purpose of this study is to test whether an individual coaching program called Social Engage Coaching (or 'Engage Coaching' for short) helps adults age 60 and older feel more connected to other people in ways that matter to them. Procedures include participating in a Social Engage Coaching program, research assessments with surveys, and assessments completed on a cell phone. Engage Coaching involves individual sessions with a trained Engage Coach (up to 10 sessions) that are designed to help participants improve social relationships and well-being. All subjects will receive the scheduled baseline and follow-up interviews by the research team. These interviews will be conducted at study start, mid-way through the program at 8 weeks and after completing the program at 16 weeks. Interviews will be via Zoom/phone as well as surveys done online.

DETAILED DESCRIPTION:
The R61 phase is a single-arm trial of S-ENG plus eCAU (n=30) with 1 week of smartphone-based target assessment at baseline, 8-weeks and 16-weeks. Participants are 30 adults age 60 and older who report clinically significant loneliness and suicide ideation and reside in a senior living community (SLC). We will use ambulatory assessment via smartphones, including both active self-report (ecological momentary assessment, EMA) and passive sensing (audio recordings & GPS) to comprehensively assess indices of social connection. Subjects will complete EMA recordings using a smartphone daily following 3 personally-selected times for prompts (to enhance recall and ease of completion of assessments) for 10-days prior to starting study interventions, beginning the day after the baseline visit. Each EMA instance takes approximately 2-5 minutes to complete. EMA will be integrated with other smartphone technology to passively capture social behavior. The Electronically Activated Recorder (EAR) will passively measure social behavior (i.e., conversation frequency, duration, and valence). GPS- will track time outside the home. Subjects will be given a study smartphone designed for older adults to use during assessment periods. All subjects who successfully complete the smartphone assessment protocol at baseline will be assigned to S-ENG. S-ENG involves 10 individual coaching sessions over (up to) 4 months. S-ENG is a stepped, modular intervention that addresses barriers to action plan implementation and challenges in processing positive outcomes when exposed to socially rewarding activities. Psychoeducational materials address the importance of social connection. Subjects complete a values clarification exercise on aspects of connection most important to participants to inform personalized activities most likely to impact loneliness. Coaches are instructed to focus action plans on activities that foster social connection. The follow-up assessments at 8- and 16-weeks include baseline measures and smartphone measures.

ELIGIBILITY:
Inclusion criteria are adults age 60 or older who live in senior living communities, endorse clinically-significant loneliness and suicide ideation over the prior month. Exclusion criteria are current problem drinking, psychosis, significant cognitive impairment, and hearing problems that preclude engagement with S-ENG and research assessors.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-06-13 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Loneliness | 16-week follow-up
  PROMIS Social Isolation Short Form 4a assessed by Ecological Momentary Assessment (EMA) on smartphones
Satisfaction with Social Activities | 16-week follow-up
  PROMIS Satisfaction with Participation in Discretionary Social Activities Short Form assessed by Ecological Momentary Assessment (EMA) on smartphones
Time in conversations | 16-week follow-up
  Smartphone passive sensing of ambient audio recordings to identify amount of time in conversations with others.
Time outside the home | 16-week follow-up
  Amount of time outside the home assessed via smartphone.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will use the NIMH Data Archive (NDA) system and procedures for its Data Sharing Plan. The NDA is a secure informatics platform for scientific collaboration and data-sharing that enables the effective communication of detailed research results, tools, and supporting documentation. Investigators will deposit all raw and analyzed data from experiments involving human subjects into this infrastructure. All data will be de-identified and will be collected from subjects who have broadly consented to share their data for research use or who have consented to share their data for research, with data use limitations.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Subject-level data (individual and derived variables) will be submitted annually using standard NDA data submission deadlines of July 15th each year. Subject-level data will be submitted in the data submission cycle following data collection (for individual variables) or data generation (for derived variables). The first data submission date will be the second cycle after the grant is awarded.
Access Criteria: Access to data for research purposes will be provided through an NDA Data Access Committee (DAC). Investigators and institutions seeking data from NDA will be expected to meet data security measures and will be asked to submit a Data Use Certification, which is cosigned by the investigator and the designated Institutional Official(s) at the NIH-recognized sponsoring institution with a current Federal Wide Assurance (FWA).
URL: https://nda.nih.gov/nda/access-data-info